CLINICAL TRIAL: NCT02836275
Title: Characterization of Ovarian Masses Unable to Classify With Ultrasound Using the International Ovarian Tumor Analysis (IOTA) Simple Rules: Value of Pelvic MRI With Perfusion- and Diffusion-weighted Imaging
Brief Title: Value of MRI in the Characterization of Ovarian Masses Unable to Classify With Ultrasound Using the International Ovarian Tumor Analysis (IOTA) Simple Rules
Acronym: IOTA-MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Dirk Timmerman, Prof. Dr., KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IOTA-MRI s59142
Record Dates: First submitted 2016-07-14; First posted 2016-07-19 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Patients With a Sonographically Unclassifiable Adnexal Mass Using the IOTA Simple Rules
Keywords: Adnexal Diseases; Ovary; Ovarian Neoplasms; Ovarian Cysts; Ovarian Diseases; Ultrasonography; Ultrasonography, Doppler; Magnetic Resonance Imaging; Diffusion Magnetic Resonance Imaging; Diagnosis; Early Diagnosis; Early Detection of Cancer; Genital Neoplasms, Female; Genital Diseases, Female; Urogenital Neoplasms; Cysts; Endocrine System Diseases; Gonadal Disorders; Neoplasms; Endocrine Gland Neoplasms; International Ovarian Tumor Analysis; Simple Rules; Preoperative Evaluation; Perfusion -and Diffusion-weighted Imaging; Adnexal Masses; Ovarian Tumors
MeSH Terms: conditions — Adnexal Diseases; Ovarian Neoplasms; Ovarian Cysts; Ovarian Diseases; Disease; Genital Neoplasms, Female; Genital Diseases, Female; Urogenital Neoplasms; Cysts; Endocrine System Diseases; Gonadal Disorders; Neoplasms; Endocrine Gland Neoplasms | interventions — Diffusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perfusion and diffusion-weighted MRI (Experimental)
  Interventions: Other: Diffusion/Perfusion-weighted Magnetic Resonance Imaging

INTERVENTIONS:
Other: Diffusion/Perfusion-weighted Magnetic Resonance Imaging

SUMMARY:
Gynecological ultrasound is well known as the preferred exam to assess patients with ovarian tumors. The International Ovarian Tumor Analysis (IOTA) group developed the 'Simple Rules' to classify an ovarian tumor as benign or malignant. In about 1/5 of patients the Simple Rules give an inconclusive result and therefore a suitable second line test is necessary. Recently the ADNEXMR SCORING system was developed, this is the first Magnetic Resonance Imaging (MRI) score system that focuses on ovarian tumors.

The aim of this prospective study is to evaluate the performance of pelvic MRI examination with perfusion -and diffusion- weighted sequences and the application of the ADNEXMR SCORING system in ovarian tumors that cannot be classified by the IOTA Simple Rules (regarding the prediction of malignancy). Other aims are the determination of the malignancy rate per ADNEXMR SCORING system class, the evaluation of interobserver reproducibility and the assessment of the accuracy of the specific diagnosis based on MRI images.

The study is a multicenter prospective study. In centers where perfusion -and diffusion weighted MRI imaging is not a part of clinical routine in unclassifiable ovarian masses based on ultrasound, the study is considered to be interventional. However, in other centres, depending on the local guidelines, perfusion -and diffusion weighted MRI imaging can be standard of care. In these centres, the study can be considered to be observational.

The IOTA-MRI project is linked to the IOTA study. In this multicenter study different diagnostic ultrasound algorithms are tested prospectively in patients with an ovarian mass prior to surgery. This study allows to define a subgroup of patients in which Simple Rules are inconclusive, in other words the population eligible for inclusion in the IOTA-MRI project. We plan to include 250 patients in the IOTA-MRI study. Patients will be included consecutively, yet only after completing the informed consent. Recruitment will take 2 years of time as of the start of the individual center.

The gold standard is the histopathology diagnosis of the mass within 120 days after ultrasound evaluation. The surgical approach is chosen by the managing clinician.

DETAILED DESCRIPTION:
Ovarian cancer is a common and lethal disease for which early detection and treatment in high volume centers and by specialized clinicians is known to improve survival. Hence, accurate methods to preoperatively characterize the nature of an ovarian tumor are pivotal. The IOTA group has suggested Simple ultrasound based rules that can be used to classify adnexal masses as benign or malignant. In about 1/5 of patients the Simple Rules give an inconclusive result and therefore a suitable second line test is necessary. The benefit of using MRI in sonographically indeterminate masses has been evaluated previously. However, the ability of MRI to correctly classify tumors unclassifiable by the IOTA Simple Rules has not been examined. The group of Thomassin-Naggara et al has recently developed the ADNEXMR SCORING system, this is the first Magnetic Resonance Imaging (MRI) score system that focuses on ovarian tumors.

The primary aim of this prospective study is to evaluate the performance of pelvic MRI examination with perfusion -and diffusion- weighted sequences and the application of the ADNEXMR SCORING system in ovarian tumors that cannot be classified by the IOTA Simple Rules (regarding the prediction of malignancy). Secondary aims are the determination of the malignancy rate per ADNEXMR SCORING system class, the evaluation of interobserver reproducibility and the assessment of the accuracy of the specific diagnosis based on MRI images.

The study is a multicenter prospective study. In centers where perfusion -and diffusion weighted MRI imaging is not a part of clinical routine in unclassifiable ovarian masses based on ultrasound, the study is considered to be interventional. However, in other centres, depending on the local guidelines, perfusion -and diffusion weighted MRI imaging can be standard of care. In these centres, the study can be considered to be observational.

The IOTA-MRI project is linked to the IOTA study. In this multicenter study different diagnostic ultrasound algorithms are tested prospectively in patients with an ovarian mass prior to surgery. This study allows to define a subgroup of patients in which Simple Rules are inconclusive, in other words the population eligible for inclusion in the IOTA-MRI project. We plan to include 250 patients in the IOTA-MRI study. Patients will be included consecutively, yet only after completing the informed consent. Recruitment will take 2 years of time as of the start of the individual center.

At first, a standardized patient history will be registered, followed by a standardized transvaginal gynecological ultrasound. All variables required for the diagnostic models as well as the subjective diagnosis and certainty of diagnosis by the examiner will be collected. Quality control is provided by the fact that all examiners involved in gynecological ultrasound have completed IOTA-training and succeeded in a certification test. All data will be registered in an online Clinical Data Miner system (CDM).

In case that the results of the Simple Rules are inconclusive, and surgery is justifiable, the patient will be informed about the IOTA-MRI study. If the patient agrees to participate, the inclusion criteria are met and if there are no contra-indications, the patient will be referred to the radiology department of the same center or an affiliated center.

Second, at the radiology department, a standardized pelvic MRI examination will take place (diffusion- and perfusion- weighted sequences). All the variables that are needed for the classification of the ADNEXMR SCORING system as well as the subjective diagnosis of the radiologist, will be registered in CDM. Quality control in this part is provided by the fact that all radiologists involved in the study are certified by EURAD (EURopean ADnex mr score).

The gold standard is the histopathology diagnosis of the mass within 120 days after ultrasound evaluation. The surgical approach is chosen by the managing clinician. In case of malignancy, staging of the tumor will be reported by the International Federation of Gynecology and Obstetrics (FIGO) classification. All results will be registered in CDM.

ELIGIBILITY:
Inclusion Criteria:

* Any adult woman with an adnexal mass unclassified by gynecological ultrasound using the IOTA Simple Rules.
* Patient planned for surgery.

Exclusion Criteria:

* Any lesion with conclusive result on gynecological ultrasound using the IOTA Simple Rules.
* Cysts that are deemed to be clearly physiological and less than 3 cm in maximum diameter are not eligible for inclusion.
* No surgery performed or surgery performed >120 days after ultrasound scan.
* Denial or withdrawal of informed consent.
* Contra-indication for MRI
* Current pregnancy
* Age < 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of the ADNEXMR SCORING system in classifying adnexal masses as malignant or benign using MRI with diffusion- and perfusion-weighted sequences in masses unclassified by the IOTA Simple Rules. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 120 days after ultrasound examination.

SECONDARY OUTCOMES:
Proportion of malignant masses per level of the ADNEXMR SCORING system. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 120 days after ultrasound examination.
Interobserver reproducibility of ADNEXMR SCORING system using MRI with diffusion- and perfusion-weighted sequences by comparing lesion characterization (interpretation) and region of interest delineation on the perfusion curve. | During estimated recruitment period of 2 years.
  This will take place later using stored images.
Accuracy of the suggested specific diagnosis made on the basis of the MRI images. | During estimated recruitment period of 2 years. Gold standard is histopathology diagnosis within 120 days after ultrasound examination.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Thomassin-Naggara, MD, PhD, Study Chair — Department of Radiology, Hôpital Tenon, Paris, FRANCE; Andrea Rockall, MBBS, MRCP, FRCR, Study Chair — Imperial College London, London, UNITED KINGDOM; Tom Bourne, MD, PhD, Study Chair — Queen Charlotte's & Chelsea Hospital, Imperial College London, London, UNITED KINGDOM; Ben Van Calster, MSc, PhD, Study Chair — Department Development & Regeneration, KU Leuven, Leuven, BELGIUM; Ignace Vergote, MD, PhD, Study Chair — Department of Obstetrics and Gynecology, University Hospitals KU Leuven, Leuven, BELGIUM
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Background] Woo YL, Kyrgiou M, Bryant A, Everett T, Dickinson HO. Centralisation of services for gynaecological cancers - a Cochrane systematic review. Gynecol Oncol. 2012 Aug;126(2):286-90. doi: 10.1016/j.ygyno.2012.04.012. Epub 2012 Apr 13. PMID 22507534
- [Background] Engelen MJ, Kos HE, Willemse PH, Aalders JG, de Vries EG, Schaapveld M, Otter R, van der Zee AG. Surgery by consultant gynecologic oncologists improves survival in patients with ovarian carcinoma. Cancer. 2006 Feb 1;106(3):589-98. doi: 10.1002/cncr.21616. PMID 16369985
- [Background] Vernooij F, Heintz AP, Witteveen PO, van der Heiden-van der Loo M, Coebergh JW, van der Graaf Y. Specialized care and survival of ovarian cancer patients in The Netherlands: nationwide cohort study. J Natl Cancer Inst. 2008 Mar 19;100(6):399-406. doi: 10.1093/jnci/djn033. Epub 2008 Mar 11. PMID 18334710
- [Background] Earle CC, Schrag D, Neville BA, Yabroff KR, Topor M, Fahey A, Trimble EL, Bodurka DC, Bristow RE, Carney M, Warren JL. Effect of surgeon specialty on processes of care and outcomes for ovarian cancer patients. J Natl Cancer Inst. 2006 Feb 1;98(3):172-80. doi: 10.1093/jnci/djj019. PMID 16449677
- [Background] Timmerman D, Testa AC, Bourne T, Ameye L, Jurkovic D, Van Holsbeke C, Paladini D, Van Calster B, Vergote I, Van Huffel S, Valentin L. Simple ultrasound-based rules for the diagnosis of ovarian cancer. Ultrasound Obstet Gynecol. 2008 Jun;31(6):681-90. doi: 10.1002/uog.5365. PMID 18504770
- [Background] Bernardin L, Dilks P, Liyanage S, Miquel ME, Sahdev A, Rockall A. Effectiveness of semi-quantitative multiphase dynamic contrast-enhanced MRI as a predictor of malignancy in complex adnexal masses: radiological and pathological correlation. Eur Radiol. 2012 Apr;22(4):880-90. doi: 10.1007/s00330-011-2331-z. Epub 2011 Nov 18. PMID 22095438
- [Background] Kinkel K, Lu Y, Mehdizade A, Pelte MF, Hricak H. Indeterminate ovarian mass at US: incremental value of second imaging test for characterization--meta-analysis and Bayesian analysis. Radiology. 2005 Jul;236(1):85-94. doi: 10.1148/radiol.2361041618. Epub 2005 Jun 13. PMID 15955864
- [Background] Thomassin-Naggara I, Aubert E, Rockall A, Jalaguier-Coudray A, Rouzier R, Darai E, Bazot M. Adnexal masses: development and preliminary validation of an MR imaging scoring system. Radiology. 2013 May;267(2):432-43. doi: 10.1148/radiol.13121161. Epub 2013 Mar 6. PMID 23468574
- [Background] Thomassin-Naggara I, Toussaint I, Perrot N, Rouzier R, Cuenod CA, Bazot M, Darai E. Characterization of complex adnexal masses: value of adding perfusion- and diffusion-weighted MR imaging to conventional MR imaging. Radiology. 2011 Mar;258(3):793-803. doi: 10.1148/radiol.10100751. Epub 2010 Dec 30. PMID 21193596
- [Background] Installe AJ, Van den Bosch T, De Moor B, Timmerman D. Clinical data miner: an electronic case report form system with integrated data preprocessing and machine-learning libraries supporting clinical diagnostic model research. JMIR Med Inform. 2014 Oct 20;2(2):e28. doi: 10.2196/medinform.3251. PMID 25600863
- [Background] Heintz AP, Odicino F, Maisonneuve P, Quinn MA, Benedet JL, Creasman WT, Ngan HY, Pecorelli S, Beller U. Carcinoma of the ovary. FIGO 26th Annual Report on the Results of Treatment in Gynecological Cancer. Int J Gynaecol Obstet. 2006 Nov;95 Suppl 1:S161-92. doi: 10.1016/S0020-7292(06)60033-7. No abstract available. PMID 17161157